CLINICAL TRIAL: NCT05306444
Title: A Phase 1 Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of CLN-418 in Subjects With Advanced Solid Tumors
Brief Title: CLN-418 Study on Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harbour BioMed US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN-418-001
Record Dates: First submitted 2022-02-24; First posted 2022-04-01 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Dose escalation (Part 1) followed by Dose expansion (Part 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CLN-418: Part 1 (Experimental): Experimental Part 1: Dose escalation
  Intravenous IV administrations of CLN-418 on Day 1 of each 21 day treatment cycle
  Dose for cohorts to be confirmed following consultation and approval by Safety Review Committee
  Interventions: Drug: CLN-418
- CLN-418: Part 2 (Experimental): Experimental Part 2: Dose Expansion
  Treatment administered at Maximum Tolerated Dose (MTD) and / or Recommended Phase 2 Dose (RP2D) established in Part 1
  Interventions: Drug: CLN-418

INTERVENTIONS:
Drug: CLN-418 — Intravenous (IV) administration
  Other Names: HBM7008

SUMMARY:
Study to evaluate the safety and tolerability of the study drug CLN-418, to determine the maximum tolerated dose and/or recommended Phase 2 study dose of CLN-418.

DETAILED DESCRIPTION:
This is a study to evaluate the safety and tolerability of the study drug CLN-418, and to determine the maximum tolerated dose and/or recommended Phase 2 study dose of CLN-418.

The study will also look at the anti-tumor activity, pharmacokinetics and immunogenicity of CLN-418.The study consists of 2 parts. In Part 1, patients are enrolled into different cohort doses in order to identify the appropriate recommended phase 2 dose (RP2D) or maximum tolerated dose (MTD). In Part 2, participants with metastatic / unresectable Non small cell lung cancer (NSCLC), Triple Negative Breast Cancer (TNBC) will receive the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) established in Part 1 of the study. In Part 1 and Part 2, participants will be administered treatment every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to sign a written informed consent document.
2. Male or female subject aged ≥18 years old at the time of screening.
3. Histologically or cytologically confirmed advanced solid tumors (e.g., breast cancer, ovarian cancer, endometrial cancer, cervical cancer, squamous cell non-small cell lung cancer (sNSCLC), cholangiocarcinoma, esophagus cancer, urothelial carcinoma, head and neck squamous cell carcinoma (HNSCC)), followed by dose-expansion cohorts (Part 2) of subjects with advanced and/or metastatic non-small cell lung cancer (NSCLC), triple-negative breast cancer (TNBC).or recurrent and progressed since last antitumor therapy for which no alternative, curative standard therapy exists.
4. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Prior used anti-B7H4 and/or anti-4-1BB antibody treatment.
2. Immuno-oncology therapy or targeted anti-cancer therapy within 4 weeks prior to first dose of investigational product, any other anti-cancer therapy within 2 weeks prior to first dose of investigational product.
3. Not yet recovered from surgery or (immune-related) toxicity related with previous treatment.
4. Known history or active infection of hepatitis B or C.
5. History of cirrhosis or non-alcohol steatohepatitis, alcohol or drug-related, autoimmune hepatitis.
6. Known brain metastases or other central nervous system metastases that are either symptomatic or untreated that require concurrent treatment.
7. Active infection that requires treatment with antibiotics or antiviral treatment within 3 weeks prior to first dose of investigational product.
8. Known history of infection with human immunodeficiency virus or known acquired immunodeficiency syndrome (AIDS).
9. Known autoimmune disease.
10. Clinically significant cardiac condition.
11. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with dose-limiting toxicity (DLT) | From Day 1 until day 21
  Number of subjects who experienced DLT events during 21 days after first administration of CLN-418, divided by the number of DLT evaluable Subjects

SECONDARY OUTCOMES:
Adverse events (AEs) according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | From signing of Informed Consent Form (ICF) till 84 days after last dose
  Number of participants with Adverse Events (including vital signs, physical examinations, and abnormal laboratory parameters).
Objective response rate, defined as the proportion of subjects with best overall response of complete response (CR) or partial response (PR) per RECIST 1.1 | From time of consent until the first documented disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefits, death or study termination whichever comes first, assessed up to 12 months
  Proportion of subjects with best overall response of complete response (CR) or partial response (PR) per RECIST 1.1
Duration of response | From time of consent until the first documented disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefits, death or study termination whichever comes first, assessed up to 12 months
  The time interval from first occurrence of a documented objective response to the time of disease progression as determined by the Investigator using RECIST 1.1 or death from any cause, whichever comes first.
Disease control rate | From time of consent until the first documented disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefits, death or study termination whichever comes first, assessed up to 12 months.
  The proportion of subjects with a best overall response of Complete Response (CR), Partial Response (PR), or stable disease (SD).
Duration of disease control | From time of consent until the first documented disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefits, death or study termination whichever comes first, assessed up to 12 months.
  The time from the date of start of treatment to the date of disease progression or death for subjects who had CR or PR or SD during treatment
Maximal tumor shrinkage | From time of consent until the first documented disease progression, unacceptable toxicity, withdrawal of consent, lack of treatment benefits, death or study termination whichever comes first, assessed up to 12 months
  The greatest tumor shrinkage achieved at any follow-up assessment
Pharmacokinetics Analysis - Serum Concentration | Up to 84 days post last dose
  Reporting of serum concentration of CLN-418
Anti-drug antibodies | Up to 84 days post last dose
  Measure of detectable Anti-drug antibody (ADA) and neutralizing antibodies in serum samples at specific study timepoints
Pharmacokinetics Analysis - Time Deviation | Up to 84 days post last dose
  Reporting time deviation data of CLN-418

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Carolina BioOncology Institute - Cancer Research Centre, Huntersville, North Carolina
  - MD Anderson, Houston, Texas
  - NEXT Oncology, Irving, Texas
- Australia (2):
  - St George Private Hospital, Kogarah, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales

IPD SHARING:
Plan to Share IPD: No
Data generated by this study will be considered confidential by the Investigator, except to the extent that it is included in a publication. The general strategy regarding publication of the study will be mutually agreed upon by the Investigator and Sponsor. The Sponsor reserves the right to manage the publication of all study results. The Investigator agrees that oral and written communication to third parties of any procedures or results from the study is subject to prior written consent of the Sponsor. Presentation material and/or manuscript(s) for publication will be reviewed by the Sponsor prior to submission for publication. Alterations in the material will only be made in agreement between the Investigator and the Sponsor